CLINICAL TRIAL: NCT05031273
Title: Designing Communities to Support Healthy Living in Aging Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1819-HQ-000051
Record Dates: First submitted 2021-06-29; First posted 2021-09-01 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy Aging
Keywords: Social connections; Healthy eating; Physical activity; Built environment; Older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The intervention arm will be exposed to the built environment intervention, and the control arm will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Residents moving into a congregate-living development with more features that support healthy living (Experimental): Residents moving into a congregate-living development designed for older adults with more design and amenities features in the building, site, and/or neighbourhood that support physical activity, healthy eating, and social connections.
  Interventions: Behavioral: Residents moving into a congregate-living development with more features that support healthy living
- Residents living in a standard congregate-living development (No Intervention): Residents living in a standard community-based congregate-living development designed for older adults.

INTERVENTIONS:
Behavioral: Residents moving into a congregate-living development with more features that support healthy living — Our team is making evidence-based recommendations to the developer and design team of an upcoming congregate-living development to support the physical activity, healthy eating, and social connections of residents moving into the new building(s). We hope for the developer to integrate into the new building(s) as many as possible of our team's built environment design and amenity recommendations into their site and/or building plans. Additionally, discussions with the municipality are also occuring on built environment design and amenity recommendations to improve the neighbourhood surrounding the site. Although our team has provided these recommendations, it is ulimatily up to the discretion of the developer and the municipality as to whether and what design and amenity changes are made.
  Arms: Residents moving into a congregate-living development with more features that support healthy living

SUMMARY:
The Housing for Health team is making evidence-based recommendations to the developer and design team of an upcoming congregate-living development to support the healthy living of older adults who will be moving into the new building. There may also be opportunities to improve the surrounding neighbourhood by collaborating with the municipality where the development is located. We will evaluate whether the intervention leads to changes in the perceived, micro-scale, and macro-scale physical built environment (BE), and whether there are impacts on the physical activity (PA), healthy eating, and social connections of residents. In parallel, we will gather qualitative data to provide a more in-depth understanding of how the BE may facilitate or hinder resident's healthy living behaviours.

DETAILED DESCRIPTION:
Background: The Housing for Health team is making evidence-based recommendations to the developer and design team of an upcoming congregate-living development to support the healthy living of older adults who will be moving into the new building. There may also be opportunities to improve the surrounding neighbourhood by collaborating with the municipality where the development is located. We will evaluate whether the intervention leads to changes in the perceived, micro-scale, and macro-scale physical built environment (BE), and whether there are impacts on the physical activity (PA), healthy eating, and social connections of residents. In parallel, we will gather qualitative data to provide a more in-depth understanding of how the BE may facilitate or hinder resident's healthy living behaviours.

Methods: This project employs a quasi-experimental pre-post design. The quantitative built environment (BE) evaluation includes assessments of macroscale (e.g., layout of communities) and microscale (e.g., street details and characteristics) changes as measured using Geographical Information Systems (GIS) and Microscale Audit Pedestrian Streetscapes (MAPS) audits, respectively. For the quantitative resident evaluation, residents moving into the intervention site or who currently live at a control site will be invited to participate. Study outcomes will be measured using self-report (i.e., surveys) and objective tools (i.e., accelerometers, Global Positioning System). The qualitative resident-environment component will be conducted using in-depth semi-structured interviews with building residents, family members, and stakeholders involved in the design/development and/or operation of the intervention site and others living in the developments' neighbourhoods. Participant observations will be completed in the building and neighbourhood environments of the intervention site.

Discussion: Findings will provide evidence on whether and how comprehensive changes to the BE of a building, site, and/or neighbourhood of a congregate living facility can impact PA, healthy eating, and social connections of older adults. Successful aspects of interventions will be scaled up in future work. We will disseminate findings to a broad audience including the scientific community via peer-reviewed publications, conference presentations, and discussion panels; and private, public, and non-profit sectors via reports, public presentations and/or communications via our partners and their networks.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years or older that are either moving into the intervention site(s), or living in a control site.

Exclusion Criteria:

* Residents who have been told by a health care provider that they have Alzheimer's or dementia.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Change in self-reported physical activity from baseline to 3-6-months post-move-in | baseline and 3-6-months post-move-in
  Self-reported physical activity will be adapted from the Neighborhood - International Physical Activity Questionnaire (N-IPAQ)
Change in self-reported physical activity from baseline to 9-12-months post-move-in | baseline and 9-12-months post-move-in
  Self-reported physical activity will be adapted from the Neighborhood - International Physical Activity Questionnaire (N-IPAQ)
Change in accelerometer-measured physical activity from baseline to 9-12-months post-move-in | baseline and 9-12-months post-move-in
  Accelerometer-measured physical activity will be measured using Actigraph accelerometers.
Change in accelerometer-measured physical activity from baseline to 3-6-months post-move-in | baseline and 3-6-months post-move-in
  Accelerometer-measured physical activity will be measured using Actigraph accelerometers.
Change in location-measured physical activity from baseline to 3-6-months post-move-in | baseline and 3-6-months post-move-in
  Location-measured physical activity will be measured using Qstarz Travel Recorder Geographical Positioning System (GPS) devices.
Change in location-measured physical activity from baseline to 9-12-months post-move-in | baseline and 9-12-months post-move-in
  Location-measured physical activity will be measured using Qstarz Travel Recorder Geographical Positioning System (GPS) devices.
Change in healthy eating from baseline to 3-6-months post-move-in | baseline and 3-6-months post-move-in
  Healthy eating will be adapted from the Nutritional Environment Measures Survey - Perceived Nutrition Environment (NEMS-P)
Change in healthy eating from baseline to 9-12-months post-move-in | baseline and 9-12-months post-move-in
  Healthy eating will be adapted from the Nutritional Environment Measures Survey - Perceived Nutrition Environment (NEMS-P)
Change in unhealthy eating from baseline to 3-6-months post-move-in | baseline and 3-6-months post-move-in
  Unhealthy eating will be adapted from the Nutritional Environment Measures Survey - Perceived Nutrition Environment (NEMS-P)
Change in unhealthy eating from baseline to 9-12-months post-move-in | baseline and 9-12-months post-move-in
  Unhealthy eating will be adapted from the Nutritional Environment Measures Survey - Perceived Nutrition Environment (NEMS-P)
Change in social connections from baseline to 3-6-months post-move-in | baseline and 3-6-months post-move-in
  Social connections will be derived from several self-report items.
Change in social connections from baseline to 9-12-months post-move-in | baseline and 9-12-months post-move-in
  Social connections will be derived from several self-report items.
Change in the micro-scale built environment from baseline to 3-6-months post-move-in | baseline and 3-6-months post-move-in
  The actual micro-scale built environment is measured using the Microscale Audit of Pedestrian Streetscapes (MAPS) audit tool
Change in the micro-scale built environment from baseline to 9-12-months post-move-in | baseline and 9-12-months post-move-in
  The actual micro-scale built environment is measured using the Microscale Audit of Pedestrian Streetscapes (MAPS) audit tool
Change in the macro-scale built environment from baseline to 3-6-months post-move-in | baseline and 3-6-months post-move-in
  The actual macro-scale built environment is measured using Geographical Information Systems (GIS)
Change in the macro-scale built environment from baseline to 9-12-months post-move-in | baseline and 9-12-months post-move-in
  The actual macro-scale built environment will be measured using Geographical Information Systems (GIS)
Change in the perceived neighbourhood built environment from baseline to 3-6-months post-move-in | baseline and 3-6-months post-move-in
  The perceived neighbourhood built environment will be measured using the Physical Activity Neighborhood Environment Scale (PANES)
Change in the perceived neighbourhood built environment from baseline to 9-12-months | baseline and 9-12-months post-move-in
  The perceived neighbourhood built environment will be measured using the Physical Activity Neighborhood Environment Scale (PANES)
Change in the perceived neighbourhood food environment from baseline to 3-6-months | baseline and 3-6-months post-move-in
  The perceived neighbourhood food environment will be measured using the Nutritional Environment Measures Survey - Perceived Nutrition Environment (NEMS-P)
Change in the perceived neighbourhood food environment from baseline to 9-12-months | baseline and 9-12-months post-move-in
  The perceived neighbourhood food environment will be measured using the Nutritional Environment Measures Survey - Perceived Nutrition Environment (NEMS-P)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stearns JA, Ren H, Spence JC, Avedzi H, Lee KK. Protocol for an evaluation of the Designing Communities to Support Healthy Living in Aging Residents Study. Arch Public Health. 2021 Oct 7;79(1):172. doi: 10.1186/s13690-021-00691-4. PMID 34620222